CLINICAL TRIAL: NCT05462431
Title: The Effect of Web-Based Deep Relaxation Exercises Applied to Pregnants on Maternal Fetal Attachment and Pregnancy Perception
Brief Title: The Effect of Web-Based Deep Relaxation Exercises in Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Nilay Gökbulut, Assist. Prof. Dr. in the Çankırı Karatekin University Midwifery Department, Çankırı Karatekin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Cankırı University
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2022-07

CONDITIONS: Maternal-Fetal Relations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- web-based deep relaxation exercise intervention (Experimental)
  Interventions: Behavioral: Deep relaxation exercises intervention
- control (No Intervention)

INTERVENTIONS:
Behavioral: Deep relaxation exercises intervention — Deep relaxation exercises intervention: breathing exercise, suitable positions for rest, and relaxation exercise instructions.
  Arms: web-based deep relaxation exercise intervention

SUMMARY:
Pregnancy is a natural but complex period in a woman's life that requires a process of adaptation to physiological, psychological and social changes. The woman first goes through a process of adaptation to pregnancy and then to motherhood. Deep Relaxation exercises, which is a low-cost and non-pharmacological method, can be effective in supporting maternal-fetal attachment and improving the perception of pregnancy. A total of 80 pregnant women (40 deep relaxation excercises and 40 control) are planned to be included in the study. Data will be collected with the 'Personel Description Form', 'Maternal Antenatal Attachment Scale (MAAS)' and 'the Pregnancy Self Perception Scale'.

DETAILED DESCRIPTION:
Pregnancy is a natural but complex period in a woman's life that requires a process of adaptation to physiological, psychological and social changes. The woman first goes through a process of adaptation to pregnancy and then to motherhood. Deep Relaxation exercises, which is a low-cost and non-pharmacological method, can be effective in supporting maternal-fetal attachment and improving the perception of pregnancy. In this study, it was aimed to determine the effect of web-based deep relaxation exercise applied to pregnant women on maternal-fetal attachment and pregnancy perception. A total of 80 pregnant women (40 deep relaxation excercises and 40 control) are planned to be included in the study. Data will be collected with the 'Personel Description Form', 'Maternal Antenatal Attachment Scale (MAAS)' and 'the Pregnancy Self Perception Scale'. A total of 80 pregnant women (40 deep relaxation excercises and 40 control) are planned to be included in the study. Data will be collected with the 'Personel Description Form', 'Maternal Antenatal Attachment Scale (MAAS)' and 'the Pregnancy Self Perception Scale'. deep relaxation excercises wiil be appliedby midwives who are experts in their fields who are certified in these fields.

ELIGIBILITY:
Inclusion Criteria:

* Having internet access,
* 24 weeks or more of pregnancy,
* There is no risk factor in pregnancy

Exclusion Criteria:

* Mental disabilities

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
Maternal Antenatal Attachment Scale (MAAS) | At the end of the 1 months
  The scale is likert type and each item is scored between 1-5. 11 items in the scale are scored in the opposite direction. There are two sub-dimensions in the scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Cankiri Karatekin University Faculty of Health Sciences, Çankırı, Centre, Turkey (Türkiye)